CLINICAL TRIAL: NCT05158192
Title: Bioavailability of a Formulation of Diosmin/Hesperidin (90/10) 500 mg Tablets With Regards to the Marketed Reference Product
Brief Title: Bioavailability of Diosmin/Hesperidin (90/10) 500 mg Tablets With Regards to Reference Product
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Andromaco S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HP8834-01
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2021-11

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Diosmin; Hesperidin; Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diosmin/Hesperidin (90/10) Test Product (Experimental): Participants received one tablet of the test formulation containing Diosmin/Hesperidin (90/10) 500 mg. The tablets was taken with water and in a fasting condition.
  Interventions: Drug: Diosmin/Hesperidin (90/10) 500 mg Test Drug
- Diosmin/Hesperidin (90/10) Reference Product (Active Comparator): Participants received one tablet of the marketed reference formulation containing Diosmin/Hesperidin (90/10) 500 mg. The tablets was taken with water and in a fasting condition.
  Interventions: Drug: Diosmin/Hesperidin (90/10) 500 mg Reference Product

INTERVENTIONS:
Drug: Diosmin/Hesperidin (90/10) 500 mg Test Drug — Investigational Medicinal Product
  Arms: Diosmin/Hesperidin (90/10) Test Product
Drug: Diosmin/Hesperidin (90/10) 500 mg Reference Product — Daflon (Trademark)
  Arms: Diosmin/Hesperidin (90/10) Reference Product

SUMMARY:
This Pilot study investigated the bioavailability in adult human subjects of 1 tablet formulations containing Diosmin/Hesperidin (90/10) 500 mg. The Pilot study was performed at a single site with 12 subjects. Participants took 1 tablets of the test product and reference product in 2 periods and 2 sequences (either test after reference or reference after test). There was a washout of 7 days between each study period.

DETAILED DESCRIPTION:
The primary objective of the study is to investigate the relative bioavailability of

Diosmin/Hesperidin (90/10) of 1 tablet formulations with Diosmin/Hesperidin (90/10) 500 mg to demonstrate bioequivalence of both formulations in terms of rate and extent of absorption:

* Test Product: Product manufactured by Laboratorios Andrómaco S.A.
* Reference Product: Daflon [Trademark], product of Les Laboratoires Servier, France.

The 90% confidence intervals for the intra-subject coefficient of variation (Test versus Reference Product) for the main pharmacokinetic parameters area under the plasma concentration-time curve from time zero to time t (AUC0-t) and from time zero to infinite (AUC0-inf), and maximum plasma concentration (Cmax) for total metabolite Diosmetin and Hesperetin was determined. Participants were confined in the study site for approximately 42 hours during each study period (for 10 hours pre-dosing and for 32 hours post dosing) during which pharmacokinetic (PK) blood samples were obtained. 21 blood samples were taken up to 32 hours after the administration in each period. Participants returned to the site to provide additional blood samples at 48 h, and 72 h postdose. The washout period between the two study periods was 7days. The samples from each participant were analyzed with validated LC-MS/MS method used for estimation of Diosmetin and Hesperetin in plasma.

The safety objective was to evaluate the tolerability of both formulations in subjects by collecting adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and/or non-pregnant, non-breast feeding female literate volunteers of 18 to 45 years (both years inclusive) with BMI of 18.50 - 29.99 Kg/m2 and weight > 50 Kg.
2. Healthy volunteers as evaluated by medical history, vitals and general clinical examination.
3. Normal or clinically insignificant biochemical, hematological, urine and serology parameters.
4. Normal or clinically insignificant ECG.
5. Negative urine test for drugs of abuse for both males and females and negative pregnancy test for females and do not plan to become pregnant during course of the study and for 03 months after completion of study.
6. Volunteers who are willing to use acceptable methods of contraception (barrier method/IUD/surgical) or abstinence, for the entire duration of the study and do not plan to be pregnant for atleast 1 month after the last drug administration.
7. Volunteers who can give written informed consent and communicate effectively.

Exclusion Criteria:

1. History of any major surgical procedure in the past 03 months.
2. History of any clinically significant cardiac, gastrointestinal, respiratory, hepatic, renal, endocrine, neurological, metabolic, psychiatric and hematological disorders.
3. History of chronic alcoholism/ chronic smoking/ drug of abuse.
4. Volunteers with known hypersensitivity to Diosmin/Hesperidin or any of the excipients.
5. History of consumption of tobacco containing products within 48 hours prior to proposed time of dosing
6. Volunteers who are positive for hepatitis B surface antigen, anti-hepatitis C antibody, treponemal antibodies and human immunodeficiency virus (HIV 1&2) antibodies.
7. Present or past history of intake of drugs or any prescription drug or over the counter (OTC) drugs within 14 days which potentially modify kinetics / dynamics of Diosmin/Hesperidin or any other medication judged to be clinically significant by the investigator.
8. History of consumption of grapefruit and/or its products within 10 days prior to the start of study.
9. Volunteers who had participated in any other clinical study or who had bled during the last 03 months before check-in.
10. History of consumption of one or more of the below, 48 hours prior to dosing: Xanthine containing food or drinks such as cola, chocolate, coffee or tea, citrus fruits or items (lime, lemon and orange), alcohol and any other food/beverage known to have interactions as deemed by the investigator
11. Volunteers who are dysphagic.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Total Diosmin/Hesperidin (90/10): area under the plasma concentration-time curve from 0 to 72 hours (AUC0-72) | From tablet intake and up to 72 hours after tablet intake
  23 samples up to 72 hours will be taken after the administration in each period.
Total Diosmin/Hesperidin (90/10): area under the plasma concentration-time curve from 0 to t hours (AUC0-t) | From tablet intake and up to 72 hours after tablet intake
  23 samples up to 72 hours will be taken after the administration in each period.
Total Diosmin/Hesperidin (90/10): Maximum plasma concentration (Cmax) | From tablet intake and up to 72 hours after tablet intake
  23 samples up to 72 hours will be taken after the administration in each period.

CONTACTS AND LOCATIONS:
Locations (1):
- Azidus Laboratories Ltd., Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No